CLINICAL TRIAL: NCT04616053
Title: A Randomised Controlled Trial to Evaluate the Effectiveness of a Multidisciplinary Team Intervention on Glycaemic Control for Disadvantaged Type 2 Diabetes Patients in France.
Brief Title: IMPACT Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pole de Sante Chambery Nord (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-A02905-34
Record Dates: First submitted 2020-10-27; First posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: primary health care; patient-centered care; poverty areas; vulnerable populations; Glycated Hemoglobin A
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): IMPACT intervention
  Interventions: Behavioral: IMPACT intervention
- Control group (No Intervention): Usual care

INTERVENTIONS:
Behavioral: IMPACT intervention — A referent is assigned to the patient. A referent is a health worker (nurse, nutritionist, psychologist …). Patient builds with his referent a free care program (without condition or limit). The patient can choose individual consultation (for example : nutrition, tabacology, psychology …) and/or collective care (for example : patient education, physical activity, relaxation …). A community health worker can help patient with his health administrative procedures. This intervention lasts 6 months.
  Arms: Intervention group

SUMMARY:
Introduction :

The prevalence of type 2 diabetes is increasing in France, especially in deprived districts.

The Itineraires Medico-sociaux Programme d'Accompagnement sur un Territoire (IMPACT) intervention is intended for disadvantaged patients with a chronic disease (not only type 2 diabetes).

The IMPACT intervention offers coordinated and patient-centered care by a multidisciplinary team with an empowerment approach. This personalised intervention lasts 6 months.

This study aims to evaluate the effect of 6 months IMPACT intervention on glycaemic control (glycated haemoglobin - HbA1c) of patients with type 2 diabetes in deprived districts.

Method :

This will be a randomised, controlled, parallel group, multicenter, open-label trial. 140 adults with type 2 diabetes will be randomised in two arms : IMPACT intervention group (n : 70) and usual care group (n : 70). The primary outcome is change in glycated haemoglobin (HbA1c) from baseline to 6 months. The primary outcome will be analysed using a linear mixed effects model.

DETAILED DESCRIPTION:
This will be a randomised, controlled, parallel group, multicenter, open-label trial. Patients will be recruited among patients with type 2 diabetes referred to the IMPACT intervention.

144 patients will be randomised in two arms : IMPACT intervention group (n : 72) and usual care group (n : 72).

IMPACT intervention : a referent is assigned to the patient. A referent is a health worker (nurse, nutritionist, psychologist …). Patient builds with his referent a free care program. The patient can choose individual consultation (for example : nutrition, tabacology, psychology …) and/or collective care (for example : patient education, physical activity, relaxation …). A community health worker can help patients with his health administrative procedures.

Patients will have 3 visits. First visit (inclusion visit) : investigator collects baseline characteristics (sociodemographic data, comorbidity, treatment, diabetes complications, weight, height, body mass index, impedancemetry, HbA1c, lipids, creatinine, albuminuria/creatinuria ratio). Then the patient will be randomised.

Second visit (midpoint visit) : investigator collects weight, BMI, impedancemetry, HbA1c and adverse events Third visit (end point visit) : investigator collects weight, BMI, impedancemetry, HbA1c, lipids and adverse events.

Analysis : The primary outcome is change in glycated haemoglobin (HbA1c) from baseline to 6 months. The primary outcome will be analysed using a linear mixed effects model. Study groups, districts, time, group-time interaction and district-group interaction will be included as fixed effects. The model will include patients as a random effect. Sub-group analysis will be made with baseline HbA1c, sex, age, Epices score (French precarity score) and diabetes duration. The robustness of the model will be tested by replacing missing data with multiple imputation methods. The same statistical modelling approach will be used for the secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes
* Inclusion HbA1c > 7.5%
* Live in Hauts de Chambéry, Biollay or Renaudie district
* Be able to give written consent

Exclusion Criteria:

* Severe cognitive or psychological disorder that may affect study understanding
* Pregnant or breastfeeding women
* Had IMPACT intervention in the previous 24 months
* Concurrent participation in another study
* Concurrent participation in another diabetes educational care program
* Life expectancy less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
HbA1c | From baseline to 6 months
  Change in glycated haemoglobin (HbA1c)

SECONDARY OUTCOMES:
HbA1c | From baseline to 3 months
  Change in glycated haemoglobin (HbA1c)
Weight | At Months 3 and 6 from baseline
  Change in weight
Body mass index | At Months 3 and 6 from baseline
  Change in body mass index
Body fat mass (Bioelectrical impedance analysis) | At Months 3 and 6 from baseline
  Change in body fat mass
Body fat percentage (Bioelectrical impedance analysis) | At Months 3 and 6 from baseline
  Change in body fat percentage
Muscle mass (Bioelectrical impedance analysis) | At Months 3 and 6 from baseline
  Change in muscle mass.
Lipids - HDL cholesterol | From baseline to 6 months
  Change in HDL cholesterol
Lipids - LDL cholesterol | From baseline to 6 months
  Change in LDL cholesterol
Lipids - triglycerides | From baseline to 6 months
  Change in triglycerides

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tricco AC, Ivers NM, Grimshaw JM, Moher D, Turner L, Galipeau J, Halperin I, Vachon B, Ramsay T, Manns B, Tonelli M, Shojania K. Effectiveness of quality improvement strategies on the management of diabetes: a systematic review and meta-analysis. Lancet. 2012 Jun 16;379(9833):2252-61. doi: 10.1016/S0140-6736(12)60480-2. Epub 2012 Jun 9. PMID 22683130
- [Background] Attridge M, Creamer J, Ramsden M, Cannings-John R, Hawthorne K. Culturally appropriate health education for people in ethnic minority groups with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2014 Sep 4;2014(9):CD006424. doi: 10.1002/14651858.CD006424.pub3. PMID 25188210
- [Background] Captieux M, Pearce G, Parke HL, Epiphaniou E, Wild S, Taylor SJC, Pinnock H. Supported self-management for people with type 2 diabetes: a meta-review of quantitative systematic reviews. BMJ Open. 2018 Dec 14;8(12):e024262. doi: 10.1136/bmjopen-2018-024262. PMID 30552277